CLINICAL TRIAL: NCT03051022
Title: The Comparison Between Dexamethasone and Morphine as an Adjuvant to Epidural Bupivacaine for Post-operative Analgesia in Lower Extremity Surgery
Brief Title: Comparison Between Dexamethasone and Morphine as an Adjuvant to Bupivacaine for Post-operative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Aida Rosita Tantri SpAn-KA, Consultant, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes008
Record Dates: First submitted 2017-02-05; First posted 2017-02-13 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Lower Extremities Fracture
Keywords: Bupivacaine; adjuvant; regional anesthesia; dexamethasone; morphine
MeSH Terms: interventions — Dexamethasone; Sodium Chloride; Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Dexamethasone 8 mg (Active Comparator): Bupivacaine 0,125% 12,5 mg combined with dexamethasone 8 mg plus NaCl 0,9% until the volume was 10 cc, prepared in a 10 cc syringe.
  Interventions: Drug: Dexamethasone 8 mg
- Morphine 2 mg (Active Comparator): Bupivacaine 0,125% 12,5 mg combined with morphine 2 mg plus NaCl 0,9% until the volume was 10 cc, prepared in a 10 cc syringe.
  Interventions: Drug: Morphine 2 mg

INTERVENTIONS:
Drug: Dexamethasone 8 mg — Dexamethasone 8 mg was given via epidural catheter as an adjuvant to 12.5 mg of 0.125% bupivacaine in 10 cc syringe and added with 0.9% sodium chloride until the volume was 10 cc.
  Other Names: 0.9 % sodium chloride, 12.5 mg of 0.125% bupivacaine
  Arms: Dexamethasone 8 mg
Drug: Morphine 2 mg — Morphine 2 mg was given via epidural catheter as an adjuvant to 12.5 mg of 0.125% bupivacaine in 10 cc syringe and added with 0.9% sodium chloride until the volume was 10 cc.
  Other Names: 0.9% sodium chloride, 12.5 mg of 0.125% bupivacaine
  Arms: Morphine 2 mg

SUMMARY:
The study aimed to compare the effectivity of dexamethasone 8 mg and morphine 2 mg as an adjuvant to epidural bupivacaine 0,125% 12,5mg for post-operative analgesia in lower extremities.

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine University of Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study and randomized into two groups. Intravenous (IV) cannula with Ringer Lactate fluid, non-invasive blood pressure monitor, electrocardiogram (ECG) and pulse-oxymetry were set on the subjects in the operation room. Epidural catheter was inserted (4 cm depth inside the epidural space) with 1,5-2 mg IV midazolam and 50 mcg IV fentanyl as premedication. The catheter insertion was confirmed with vacuum aspiration and negative test-dose. General anesthesia induction was done by fentanyl 2 mcg/kg, propofol 2 mg/kg, and atracurium 0,5 mg/kg. Maintenance was done by sevoflurane 2vol%, fentanyl and atracurium. Surgery starts without intraoperative epidural regimen. Surgery duration, blood pressure, heart rate, respiratory rate, oxygen saturation by pulse oximetry (SpO2) were recorded. For post-operative analgesia, subjects received paracetamol 1 gr IV and intermittent epidural analgesia regimen in a 10 cc syringe: Group 1 received Bupivacaine 0,125% 12,5 mg combined with dexamethasone 8 mg plus 0,9% sodium chloride (NaCl) until the volume was 10 cc; Group 2 received Bupivacaine 0,125% 12,5 mg combined with morphine 2 mg plus 0,9% NaCl until the volume was 10 cc. The injection was given by anesthesiology residents without knowing the syringe's content. Patient Controlled Analgesia (PCA) morphine was given in the recovery room. Data recorded were blood pressure, heart rate, respiratory rate, oxygen saturation, visual analog scale, side effects, the time when first additional analgesia was needed by subjects, the opioid requirement within 24 hours post-operation. Data was analyzed using Statistical Package for the Social Sciences (SPSS) software, for numerical data using unpaired T-test or Mann-Whitney-U test, for categorical data using Chi-square or Fisher Exact Test. Data normality was tested by Kolmogorov-Smirnov test. Significant value is p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-60 years old with American Society of Anesthesiologists (ASA) physical status I-II and body mass index (BMI) 18,5-25 kg/m2 who were planned to undergo lower extremity surgery
* Subjects have been explained about the study, have agreed to enroll and have signed the informed consent form

Exclusion Criteria:

* Subjects with history of bupivacaine allergy
* Subjects with history of morphine allergy
* Subjects with history of urine retention
* Subjects with history of gait disturbance or using prosthetic, Subjects with history of peptic ulcer
* Subjects with history of long term use of corticosteroid
* Subjects with contraindications for epidural anesthesia
* Subjects rejected to participate in the study.

Drop out criteria:

* Subjects with epidural anesthesia complications (e.g. shock, anaphylactic reaction, seizures, severe respiratory disturbance)
* Subjects with failed epidural anesthesia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
The degree of pain at 24-hours post-operative | 24 hours post-operative
  The degree of pain was measured using Visual Analog Scale (VAS)
The time for first requested post-operative additional analgesia | 24 hours post-operative
  How long (in minutes) until the subject requested for an additional analgesics after surgery.
The opioid requirement with the first 24-hours post-operative | 24-hours post-operative
  Patient Controlled Analgesia (PCA) measured the opioid requirement in milligram.

SECONDARY OUTCOMES:
Side Effects | 24-hours post-operative
  Side effects measured were incidences of nausea/vomiting, motoric inhibition, sedation, respiratory depression, hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Aida R Tantri, PhD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Central Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pakzad H, Roffey DM, Knight H, Dagenais S, Yelle JD, Wai EK. Delay in operative stabilization of spine fractures in multitrauma patients without neurologic injuries: effects on outcomes. Can J Surg. 2011 Aug;54(4):270-6. doi: 10.1503/cjs.008810. PMID 21651838
- [Background] Nicola R. Early Total Care versus Damage Control: Current Concepts in the Orthopedic Care of Polytrauma Patients. ISRN Orthop. 2013 Mar 21;2013:329452. doi: 10.1155/2013/329452. eCollection 2013. PMID 24959356
- [Background] Xing D, Chen Y, Ma JX, Song DH, Wang J, Yang Y, Feng R, Lu J, Ma XL. A methodological systematic review of early versus late stabilization of thoracolumbar spine fractures. Eur Spine J. 2013 Oct;22(10):2157-66. doi: 10.1007/s00586-012-2624-1. Epub 2012 Dec 22. PMID 23263169
- [Background] Ramsay MA. Acute postoperative pain management. Proc (Bayl Univ Med Cent). 2000 Jul;13(3):244-7. doi: 10.1080/08998280.2000.11927683. No abstract available. PMID 16389390
- [Background] Voscopoulos C, Lema M. When does acute pain become chronic? Br J Anaesth. 2010 Dec;105 Suppl 1:i69-85. doi: 10.1093/bja/aeq323. PMID 21148657
- [Background] Garimella V, Cellini C. Postoperative pain control. Clin Colon Rectal Surg. 2013 Sep;26(3):191-6. doi: 10.1055/s-0033-1351138. PMID 24436674
- [Background] Moraca RJ, Sheldon DG, Thirlby RC. The role of epidural anesthesia and analgesia in surgical practice. Ann Surg. 2003 Nov;238(5):663-73. doi: 10.1097/01.sla.0000094300.36689.ad. PMID 14578727
- [Background] Becker DE, Reed KL. Essentials of local anesthetic pharmacology. Anesth Prog. 2006 Fall;53(3):98-108; quiz 109-10. doi: 10.2344/0003-3006(2006)53[98:EOLAP]2.0.CO;2. PMID 17175824
- [Background] Becker DE, Reed KL. Local anesthetics: review of pharmacological considerations. Anesth Prog. 2012 Summer;59(2):90-101; quiz 102-3. doi: 10.2344/0003-3006-59.2.90. PMID 22822998
- [Background] Mercanoglu E, Alanoglu Z, Ekmekci P, Demiralp S, Alkis N. Comparison of intravenous morphine, epidural morphine with/ without bupivacaine or ropivacaine in post-thoracotomy pain management with patient controlled analgesia technique. Braz J Anesthesiol. 2013 Mar-Apr;63(2):213-9. doi: 10.1016/S0034-7094(13)70218-6. PMID 23601264
- [Background] Nordquist D, Halaszynski TM. Perioperative multimodal anesthesia using regional techniques in the aging surgical patient. Pain Res Treat. 2014;2014:902174. doi: 10.1155/2014/902174. Epub 2014 Jan 20. PMID 24579048
- [Background] Tomar GS, Godwin RB, Gaur N, Sethi A, Narang N, Kachhwaha V, Kriplani TC, Tiwari A. A double-blind study on analgesic effects of fentanyl combined with bupivacaine for extradural labor analgesia. Anesth Essays Res. 2011 Jul-Dec;5(2):147-52. doi: 10.4103/0259-1162.94754. PMID 25885378
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Background] Gan TJ, Meyer T, Apfel CC, Chung F, Davis PJ, Eubanks S, Kovac A, Philip BK, Sessler DI, Temo J, Tramer MR, Watcha M; Department of Anesthesiology, Duke University Medical Center. Consensus guidelines for managing postoperative nausea and vomiting. Anesth Analg. 2003 Jul;97(1):62-71, table of contents. doi: 10.1213/01.ane.0000068580.00245.95. PMID 12818945
- [Background] Hefni AF, Mahmoud MS, Al Alim AA. Epidural dexamethasone for post-operative analgesia in patients undergoing abdominal hysterectomy: A dose ranging and safety evaluation study. Saudi J Anaesth. 2014 Jul;8(3):323-7. doi: 10.4103/1658-354X.136420. PMID 25191180
- [Background] Thomas S, Beevi S. Epidural dexamethasone reduces postoperative pain and analgesic requirements. Can J Anaesth. 2006 Sep;53(9):899-905. doi: 10.1007/BF03022833. PMID 16960268